CLINICAL TRIAL: NCT02613260
Title: Mailed FIT Outreach to Improve Colon Cancer Screening in the Safety-net System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Stanford University (Other); San Francisco Department of Public Health (Other Government)
Responsible Party: Principal Investigator, Ma Somsouk, MD, MAS, Associate Professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14-14861
Record Dates: First submitted 2015-11-20; First posted 2015-11-24 (Estimated); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Colonic Neoplasms
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): Patients in this study arm will receive usual care from their primary care clinic.
- FIT Outreach + Usual Care (Experimental): Patients in this study arm will receive usual care at their primary care clinic and the intervention.
  Interventions: Behavioral: FIT Outreach

INTERVENTIONS:
Behavioral: FIT Outreach — This arm will consist of priming patients with a postcard and a possibly a phone call two weeks prior to them being mailed a FIT kit. The FIT kits will be mailed to the patients with a letter from their clinic's care team informing them why they should complete the FIT and wordless instructions to help them complete the FIT. Two weeks after the FIT kit is mailed the patients that have not returned the kit will receive up to two reminder calls. During the phone calls the outreach workers will use health coaching techniques to encourage patients to complete the FIT. All written materials have been translated into English and Chinese and during phone calls patients will be spoken to in the language that they are most comfortable using.
  Arms: FIT Outreach + Usual Care

SUMMARY:
Uptake of colorectal cancer (CRC) screening is suboptimal in the San Francisco Health Network and access to care may be limited so novel models of health care delivery are warranted. The objective of this study is to examine whether a centralized panel management model with mailed fecal immunochemical test (FIT) will be effective at increasing the uptake of CRC screening and could be developed and sustained within the typical parameters of cost-effectiveness and budget impact analyses.

DETAILED DESCRIPTION:
Rationale: Since uptake of colorectal cancer (CRC) screening is suboptimal in the SF safety-net system and access to care may be limited, novel models of health care delivery are warranted. The overall hypothesis is that a centralized panel management model with mailed fecal immunochemical test (FIT) will be effective at increasing the uptake of CRC screening and could be developed and sustained within the typical parameters of cost-effectiveness and budget impact analyses. Barriers to immunization of adults include missed opportunities during visits, limited access to providers, and provider and patient beliefs of efficacy.

Design: To rigorously examine the benefit of the centralized panel management to improve uptake of CRC screening with mailed FIT, the electronic health system will be used to identify eligible patients who are not up-to-date with CRC screening. Broadly, patients will be randomized 1:1 to usual care or intervention arm, stratified by clinic, gender, prior screening, and race to receive mailed FIT kits + usual care versus usual care alone. The cost-effectiveness of no screening, usual care, and centralized management with mailed FIT outreach will be compared using mathematical simulation models.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic men and women
* 50 to 75 years of age

Exclusion Criteria:

* Personal history of polyps requiring colonoscopic surveillance
* Homeless
* Severe co-morbidities limiting life expectancy e.g., advanced stage cancer

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13470 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Completion of FIT- one year | One year
  The primary outcome is the completion rate for CRC screening one-year after randomization between mailed FIT outreach and usual care.

SECONDARY OUTCOMES:
Incomplete FIT- 28 days | 28 days
  Of the patients mailed the FIT kit the number of patients that have not completed their FIT.
FIT Positive | 1 year
  Among the patients that have completed the FIT the percentage that had a positive FIT test.
Completed Colonoscopy | One year
  Of the patients that had a positive FIT the percentage of patients that received a colonoscopy.
Colonoscopy Findings | One year
  Of the patients that received a colonoscopy what were the findings (rate of any adenoma, advanced neoplasia, and colorectal cancer).
Cost | Two years
  How much the program costed to start and the costs throughout program implementation.

CONTACTS AND LOCATIONS:
Overall Officials: Ma Somsouk, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco-San Francisco General Hospital, San Francisco, California, United States

REFERENCES:
- [Derived] McClellan SP, Canchola AJ, Potter MB, Gomez SL, Somsouk M. Neighborhood socioeconomic status and the effectiveness of colorectal cancer screening outreach with mailed fecal immunochemical tests within a safety net healthcare system in San Francisco, CA: A subgroup analysis of a randomized controlled trial. Prev Med. 2023 Feb;167:107388. doi: 10.1016/j.ypmed.2022.107388. Epub 2022 Dec 14. PMID 36528113
- [Derived] Lee B, Keyes E, Rachocki C, Grimes B, Chen E, Vittinghoff E, Ladabaum U, Somsouk M. Increased Colorectal Cancer Screening Sustained with Mailed Fecal Immunochemical Test Outreach. Clin Gastroenterol Hepatol. 2022 Jun;20(6):1326-1333.e4. doi: 10.1016/j.cgh.2021.07.022. Epub 2021 Jul 16. PMID 34280552
- [Derived] Wang A, Rachocki C, Shapiro JA, Issaka RB, Somsouk M. Low Literacy Level Instructions and Reminder Calls Improve Patient Handling of Fecal Immunochemical Test Samples. Clin Gastroenterol Hepatol. 2019 Aug;17(9):1822-1828. doi: 10.1016/j.cgh.2018.11.050. Epub 2018 Nov 29. PMID 30503967